CLINICAL TRIAL: NCT06121193
Title: Using Interventional Informatics to Address Social Determinants of Health During Clinical Care Visits to Promote Behavior Change and PREVENT Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202004230
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients - Wait-List Control (Active Comparator): Complete questionnaires at baseline (administered electronically or by mail). Follow-up measures will be administered at 3-months after the clinic visit electronically and by mail.
  • A PREVENT action plan (behavior change prescription, community resources, and education) will be provided to the patient via email after the completion of the follow-up measurement.
  Interventions: Behavioral: Wait-list Control
- Experimental: Patients - PREVENT Tool (Experimental): Complete questionnaires at baseline (administered electronically or by mail). Follow-up measures will be administered immediately following the clinic visit, and monthly for 3-months after the clinic visit electronically and by mail
  • At the clinic visit, the provider will use the PREVENT tool to discuss CVH risk and deliver a tailored behavioral change plan inclusive of patient-centered community resources.
  Interventions: Behavioral: PREVENT tool
- Providers (No Intervention): -All eligible providers will be sent questionnaires electronically to their email at baseline, following provider training and follow-up. Providers will be invited to attend a training session to educate them on the PREVENT tool at baseline.

INTERVENTIONS:
Behavioral: PREVENT tool — PREVENT is a novel Health Information Technology tool designed to promote physical activity and healthy food intake among overweight/obese patients at the point of care. PREVENT automates the delivery of personalized, evidence-based behavior change recommendations and provides an interactive map of community resources to help providers link patients to resources in their community.
  Arms: Experimental: Patients - PREVENT Tool
Behavioral: Wait-list Control — Will receive routine clinical care. After completion of follow-up measures, control participants will receive a behavior change prescription via the PREVENT tool
  Arms: Patients - Wait-List Control

SUMMARY:
Healthcare providers recognize the need for behavior change and the influence of social determinants on youth at risk for poor cardiovascular health (CVH), especially among those of low-socioeconomic status (SES). Yet, providers lack the time and community data necessary to provide tailored, evidence-based care within routine practice. This project will use an Interventional Informatics approach to help providers prescribe patient-centered, evidence-based physical activity and nutrition prescriptions and link patients to community resources to account for social determinants at the point-of-care. This project will integrate our existing, novel, Patient-centered Real-timE interVENTion (PREVENT) tool into the BJC electronic health record (EHR) and test it with providers and adolescent patients at-risk for poor CVH. EHR integration of PREVENT will enable a cyclical, synergistic and data-centric approach to impact modifiable risk factors (physical activity and food intake) and prevent cardiovascular disease. This approach uses health informatics technology (HIT) to deliver data-driven, patient-centered care and generate evidence to support the use of HIT as a way to prevent cardiovascular disease across diverse patients and communities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-17 years at baseline
* at risk for poor CVH (body mass index >= 85th percentile)
* Receiving care from the Healthy Start Clinic at Barnes Jewish Hospital.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction of PREVENT tool: survey | 3-months
  A survey (6-questions) will assess patient's satisfaction with the PREVENT tool. Questions are asked on a 5-point Likert scale (range: 6-30) with a higher score indicating greater satisfaction.
Provider's satisfaction of PREVENT tool: survey | 3-months
  A survey (31-questions) will assess provider's acceptability and satisfaction with five aspects of health information technology: content, accuracy, format, ease of use and timeliness. Questions are asked on a 5-point Likert scale (range: 31-155) with a higher score indicating greater satisfaction.
Fidelity of PREVENT tool implementation | 0-3 months
  Fidelity will be measured using direct observation of patient-provider interactions while using the PREVENT tool. A direct observation checklist will be used by the observer to determine the number of interactions with the PREVENT tool that were implemented as intended.

SECONDARY OUTCOMES:
Change in patient's motivation | At baseline, and 3-months
  A survey (15-question) administered to patients will assess motivation and self-efficacy for behavior change. Questions are asked using a 4-point Likert scale (range: 15-60) with a higher score indicating greater motivation.
Change in patient's knowledge of CVH | At baseline, and 3-months
  A survey (3-question) administered to patients to assess their knowledge of CVH risk (perceived value/importance of healthy behaviors) and awareness of resources. Questions are asked using a 4-point Likert scale (range: 3-12) with a higher score indicating greater knowledge.
Change in food intake behaviors | At baseline, and 3-months
  Patient-reported food intake behaviors (fruit and vegetable intake, whole grains, sugar-sweetened beverages and snacking behaviors) are collected using a brief Health Behavior & Attitudes Survey.
Change in physical activity behaviors | At baseline, and 3-months
  Patient-reported physical activity (minutes of moderate and vigorous activity per week) are collected using a survey (4-questions). Patients report the average number of minutes of moderate and vigorous activity they do per week.
Change in body mass index z-score | At baseline, and 3-months
  Collected from patient's medical record. BMI z-score was calculated using the Centers for Disease Control and Prevention Growth Charts. The mean change was calculated by subtracting the baseline mean from the follow-up mean for each intervention group.
Change on patient's average systolic and diastolic blood pressure | At baseline, and 3-months
  Collected from patient's medical record
Change in patient's cholesterol | At baseline, and 3-months
  Collected from patient's medical record
Change in patient's blood glucose | At baseline, and 3-months
  Collected from patient's medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kepper M, Walsh-Bailey C, Miller ZM, Zhao M, Zucker K, Gacad A, Herrick C, White NH, Brownson RC, Foraker RE. The Impact of Behavior Change Counseling Delivered via a Digital Health Tool Versus Routine Care Among Adolescents With Obesity: Pilot Randomized Feasibility Study. JMIR Form Res. 2024 May 17;8:e55731. doi: 10.2196/55731. PMID 38758581